CLINICAL TRIAL: NCT02351830
Title: Controlled Birch Pollen Challenge in the Environmental Exposure Unit (EEU); Clinical Validation and Biomarker Exploration
Brief Title: Clinical Validation of Birch Pollen in the EEU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University (Other)
Collaborators: University of British Columbia (Other)
Responsible Party: Principal Investigator, Dr. Anne Ellis, Chair, Division of Allergy & Immunology, Queen's University
Other Study IDs: Birch Validation Study
Record Dates: First submitted 2015-01-27; First posted 2015-01-30 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2015-04

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic | interventions — PR-10 protein, walnut birch pollen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Birch Pollen — Participants will be exposed to birch pollen to activate their allergy symptoms therefore validating the unit.
Procedure: Nasal Brushing — To assess allergic biomarkers participants will provide a nasal sample which will be collected using a cytobrush. This procedure will be performed twice; once at screening and once following pollen exposure in the EEU.

SUMMARY:
The EEU has proven effective in multiple studies evaluating various aspects of seasonal allergic rhinitis. All previous EEU clinical trials have utilized ragweed or grass pollen as the allergen of choice for dispersal, due to the local population, but many emerging treatments for allergic rhinitis are allergen specific, thus it is desirable to expand the repertoire of pollen selection for use in the EEU. Ragweed, grass and birch pollen have differing appearances and sizes but essentially, both have characteristics which promote the ability to keep the pollen grains suspended and hence, the ability to maintain proper concentrations within the EEU. Preliminary validation studies conducted in the EEU, absent of human volunteers, have confirmed our ability to release, disperse and maintain birch pollen concentrations in the EEU using the existing technology.

This study aims to validate the use of birch pollen on a clinical scale. By adding non- allergic participants into the EEU, the investigators hope to determine if non-allergic persons exhibit differences at baseline in their "epigenetic biomarkers" from those who have pre-existing and established allergic airways inflammation.

DETAILED DESCRIPTION:
The Environmental Exposure Unit (EEU) is a controlled allergen challenge model of allergic rhinitis ('hayfever') that has been used extensively to study various anti-allergic therapies. The EEU is a unique, internationally recognized research facility that allows for the exposure of groups of as few as 5 to as many as 150 volunteers simultaneously to ambient levels of airborne allergens such as ragweed pollen and provides a unique study environment ideally suited to evaluate efficacy and onset of action of various anti-allergic medications. This specialized facility, located within Kingston General Hospital, allows for the tight regulation of environmental variables such as air quality, temperature, humidity and CO2 levels as well as the precise maintenance of allergen concentration within this specialized room. Thus the EEU provides a closed environment in which participants are exposed to a predetermined, controlled, constant level of airborne pollen. All previous studies have used either ragweed or grass pollen, and the investigators have not clinically validated the use of birch pollen in the EEU. This study will confirm that the birch pollen circulated in the EEU can generate allergic rhinitis symptoms similar to those seen in the 'real world', and will also provide an opportunity to collect blood from participants before and after allergen challenge in order to better understand allergic inflammation, to hopefully someday identify novel therapies in allergic disease.

This study will consist of a Screening Visit and one pollen exposure visit. The duration of each participant's participation in the study from Screening to End of Study (EOS) will be approximately 3 weeks. The study population will consist of healthy, ambulatory male and female volunteers, 18-65 years of age with either a history of seasonal allergic rhinitis or a history of no allergic reactions. Approximately 55-75 participants will be screened to ensure 50 eligible participants are enrolled into the study (40 allergic, 10 non-allergic).

All participants will give written informed consent prior to any study procedures being performed. Participants who meet all inclusion/exclusion criteria during the screening process will be asked to return to the EEU for their pollen exposure visit. At the Screening visit participants will provide a full medical history and undergo a physical examination. They will have their height/weight and vitals measured and skin testing will be performed to confirm allergic response to a panel of common aeroallergens (or lack of response for the non-allergic individuals). Women of child bearing potential will undergo a urine pregnancy test to rule out pregnancy. Eligible participants will be asked to return to the research site for one 4 hour exposure to birch pollen in the Environmental Exposure Unit (EEU). Peripheral blood samples will be collected before and after pollen exposure for measurement of potential biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* minimum 2 year document history of rhinoconjunctivitis during typical tree pollen season (mid March to early May) OR completely non-atopic (allergic) to all environmental allergens.
* positive skin test to birch allergen OR negative skin test to a panel of allergens at screening.

Exclusion Criteria:

* participants with asthma.
* participant is pregnant, lactating or actively trying to conceive.
* participant is currently receiving allergen specific immunotherapy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2015-01; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Change in Total Nasal Symptom Score from Baseline to each time point. | Second and Final Visit (4 hour pollen exposure)
  Participants will assess their symptoms every 30 minutes during the 4-hour pollen exposure session and the sum of the 4 nasal symptoms (runny nose, stuffy nose, sneezing and itchy nose) which create the Total Nasal Symptom Score (TNSS)

SECONDARY OUTCOMES:
Percentage of people achieving a TNSS of 6 or greater | Second and Final Visit (4 hour pollen exposure)
  The data will be evaluated to see how many participants achieved a TNSS of 6 or greater (out of a possible 12) at the second hour of pollen exposure. This is typically the time frame for qualification for randomization in a clinical trial.
Percentage of people achieving a TRSS of 10 or greater | Second and Final Visit (4 hour pollen exposure)
  The data will be evaluated to see how many participants achieved a TRSS of 10 or greater (out of a possible 24) during the second hour of pollen exposure.
Change in Total Rhinoconjunctivitis Symptom Score from Baseline to each time point. | Second and Final Visit (4 hour pollen exposure)
  Participants will assess their symptoms every 30 minutes during the 4-hour pollen exposure session and the sum of all of their symptoms (nasal symptoms listed above as well as itchy eyes, watery/tearing eyes, red burning eyes and itching of the ears/palate/throat) which create the Total Rhinoconjunctivitis Symptom Score (TRSS)
Change in Peak Nasal Expiratory Flow (PNIF) from baseline at each time point. | Second and Final Visit (4 hour pollen exposure)
  Participants will measure their nasal blockage using a Peak Nasal Inspiratory Flow meter every 30 minutes at the same time that they measure the rest of their symptoms. As the participant's nose become more congested this value should decrease.

CONTACTS AND LOCATIONS:
Overall Officials: Anne K Ellis, MD, Principal Investigator — Queen's University
Locations (1):
- Kingston General Hospital, Kingston, Ontario, Canada

REFERENCES:
- [Derived] Ellis AK, Soliman M, Steacy LM, Adams DE, Hobsbawn B, Walker TJ. Clinical validation of controlled exposure to birch pollen in the Environmental Exposure Unit (EEU). Allergy Asthma Clin Immunol. 2016 Oct 19;12:53. doi: 10.1186/s13223-016-0156-7. eCollection 2016. PMID 27777594